CLINICAL TRIAL: NCT04406519
Title: Static Postural Balance Evaluation in Children With Severe Haemophilia and Investigation of Its Relationship With Joint Health: a Cross-sectional Study
Brief Title: Evaluation of Static Postural Balance in Children With Hemophilia and Its Relationship With Joint Health
Status: Completed | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Necati Muhammed TAT, Lecturer, Necmettin Erbakan University
Other Study IDs: Necmettin Erb. Physiotherapy-3
Record Dates: First submitted 2020-05-20; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Hemophilia; Arthropathy of Knee; Arthropathy of Ankle or Foot
Keywords: haemophilia; balance; joint health; arthropathy; children
MeSH Terms: conditions — Hemophilia A; Joint Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemophilia Group: The inclusion criteria in the hemophilia group were as follows; patients aged 6 to 18 years who developed HA in at least one of the lower limb joints due to severe haemophilia (total lower limb HJHS ≥3); to be receiving prophylaxis but have no major bleeding that could affect the musculoskeletal system in the past two weeks; and who did not perform regular physical activity and sports.
- Control Group: The control group was consisted of healthy peers. The exclusion criteria in the control group were as follows: who had any auditory and visual impairment; who underwent orthopedic injuries including lower limb; and who had any neurological or cognitive impairment that could affect balance.

SUMMARY:
Hemophilia is a rare hematological disorder characterized by a partial or complete deficiency of clotting factor VIII or IX.Bleeding disorders mainly affect the musculoskeletal system. Intra-articular bleeding is an important complication related to hemophilia and usually occurs in large synovial joints such as knees and ankles. Initially, these bleeds occur non-specific spontaneously and usually affect one joint, and repeated bleeding makes that joint a target joint. Postural balance can be defined as the ability to maintain a stable posture for maximum duration with minimal body sway, or to hold the body centre of gravity (CoG) over its base support in varying conditions (1). Somatosensorial information from mechanoreceptors, visual and vestibular receptors is required to maintain postural balance. Postural balance is tried to be controlled by the postural adjustments provided by the contraction of the lower limb muscles and trunk muscles before perturbation. Spontaneous hemarthrosis is a distinctive feature of severe haemophilia, and that recurrent bleedings may likely to cause postural balance disorders by disrupting proprioceptive inputs from mechanoreceptors in the joint. Data on how bleeding affects postural balance in children with hemophilia is unclear.In the relationship between the clinical evaluation of hemophilia and postural balance, there is little research in the literature.

DETAILED DESCRIPTION:
The aim of this study was to investigate the changes in static postural balance parameters more reliably and comprehensively with a longer test duration and to reveal the relationship between balance parameters and joint health score in children with hemophilia. The investigator's hypothesis was that in children with hemophilia (CwH), postural balance was correlated with joint health status and had poor static postural balance compared to healthy peers.

Twenty-one CwH aged 6 to 18 years who developed hemophilic arthropathy in at least one of the lower limb joints due to severe hemophilia and twenty-one healthy peers were included in the study.

The Hemophilia Joint Health Score (HJHS), a valid and reliable test, was used to measure the joint health in CwH. Muscle strengths were measured with digital dynamometer. The kinetic devices most commonly used to evaluate in the laboratory evaluation of postural balance are the force platform and are considered the gold standard method. In the postural balance evaluation, changes in the X and Y axis were used. The amplitude of these changes, the standard deviation of the displacement, and the velocity were evaluated. In addition, the ellipse area and perimeter were measured.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 to 18 years
* Participants do not perform regular physical activity and sports.
* For hemophilia group who developed hemophilic arthropathy in at least one of the lower limb joints due to severe hemophilia (total lower limb hemophilia joint health score ≥3).
* For hemophilia group patients to be receiving prophylaxis but have no major bleeding that could affect the musculoskeletal system in the past two weeks

Exclusion Criteria:

* Have any auditory and visual impairment
* Undergo any orthopedic injuries including lower limb
* Have any neurological or cognitive disorders

Ages: 6 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Hemophilic children in Van province
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Hemophilia Joint Health Score | 1 month
  The score for each index-joint range from 0 to 20 and the lower limb joint score from 0 to 80. A high score indicates that the joint health is worse.
Center of Pressure (CoP)- CoPX and CoPY | 1 month
  Amplitude of CoP is the difference between the biggest and smallest CoP displacement for X-axis (CoPX) and Y-axis (CoPY), the smaller the score, the better the postural stability.
Velocity- Mediolateral (MLV) and Anteroposterior (APV) | 1 month
  The velocity is calculated by dividing the CoP excursion by trial time and expressed in mm/sec. It reflects the effectiveness of the postural stability- the bigger the velocity indicates the worse the postural control.
Standard deviation of body sway- Mediolateral (MLSD) and Anteroposterior (APSD) | 1 month
  The lower standard deviation in the body sway indicates that the postural balance is well.
Ellipse Area | 1 month
  %90 of the total area scanned in the mediolateral and anteroposterior direction is calculated using an ellipse. A high score indicates that postural balance is worse
Perimeter | 1 month
  Quantifies the size of the displacement based upon the total distance scanned in mm, and the higher the length of the scanned area considered that postural stability is poor
Muscle strength | 1 month
  The flexors and extensors of the knee were measured by giving the resistance from proximal malleoli when the hip and knee were in 90° flexion during sitting position. The dorsi and plantar flexors of ankle were measured in the lower limb stabilized in supine position, giving resistance from the proximal of the metatarsophalangeal joint and was recorded in pounds.
Standard deviation of the trunk | 1 month
  Total,anteroposterior and mediolateral standard deviation of the trunk were measured in degrees by the sensors. The lower standard deviation in the trunk sway indicates that the postural balance is well.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Fayik Oner, Prof., Study Chair — Van Yuzuncu Yil University Faculty of Medicine Dept of Pediatric Hematology; Kamuran Karaman, Assoc. Prof., Study Director — Van Yuzuncu Yil University Faculty of Medicine Dept of Pediatric Hematology; Seyhmus Kaplan, Assoc. Prof., Principal Investigator — Van Yuzuncu Yil University Faculty of Medicine Dept of Sports Medicine
Locations (1):
- Yuzuncu Yil University, Van, Bardakcı, Turkey (Türkiye)